CLINICAL TRIAL: NCT03780751
Title: Randomized-controlled Comparison of Two Online-interventions: How Effective Are Cognitive-behavioral and Mindfulness-based Sexual Therapy in Improving Sexual Desire in Women With Hypoactive Sexual Desire Disorder?
Brief Title: Waitlist Controlled Comparison of Cognitive-behavioral vs. Mindfulness-based Online-treatments for Women With Low Sexual Desire
Acronym: MiSELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Julia Velten, Postdoctoral Research Associate, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VE 1083/2-1
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: Sexual dysfunction; Female Sexual Interest/Arousal Disorder; Internet-based intervention; Mindfulness; Cognitive-behavioral therapy
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups parallel for the duration of the study. 40% of participants will be assigned to one of the two immediate treatment conditions, 20% of participants will be assigned to a waitlist and will begin active treatment after a six months waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-behavioral treatment (Experimental): COPE-program of 8 sessions (+ 1 booster session) of guided Internet-based treatment including psychoeducation, sexual education, guided masturbation, sensate focus and cognitive-behavioral interventions (e.g., thought diaries, challenging of maladaptive thought patterns, behavioral analysis). Participants are encouraged to practice exercises between sessions.
  Interventions: Behavioral: Cognitive-behavioral treatment
- Mindfulness-based treatment (Experimental): MIND-program of 8 sessions (+ 1 booster session) of guided Internet-based treatment including psychoeducation, sexual education, guided masturbation, sensate focus and mindfulness-based exercises (e.g., breathing meditation, body scan, sitting meditation).
  Interventions: Behavioral: Mindfulness-based treatment
- Waitlist (No Intervention): Participants will receive no immediate treatment but will be able to choose either MIND or COPE after a six months waiting period.

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment — COPE-program of 8 sessions (+ 1 booster session) of guided Internet-based treatment including psychoeducation, sexual education, guided masturbation, sensate focus and cognitive-behavioral interventions (e.g., thought diaries, challenging of maladaptive thought patterns, behavioral analysis). Participants are encouraged to practice exercises between sessions.
  Arms: Cognitive-behavioral treatment
Behavioral: Mindfulness-based treatment — MIND-program of 8 sessions (+ 1 booster session) of guided Internet-based treatment including psychoeducation, sexual education, guided masturbation, sensate focus and mindfulness-based exercises (e.g., breathing meditation, body scan, sitting meditation).
  Arms: Mindfulness-based treatment

SUMMARY:
Problems with sexual function are common and distressing. The most frequent sexual difficulty in women is a lack of sexual desire with a prevalence of 20-30%. When low sexual desire is experienced over several months and causes significant personal distress, a sexual dysfunction can be diagnosed (ICD-10: Hypoactive Sexual Desire Disorder: HSDD). A distressing lack of desire is reported by 6% of sexually active women. Psychological interventions are the treatment of choice for women with HSDD. Promising treatment approaches include cognitive-behavioral and mindfulness-based interventions. A recent meta-analysis also showed that Internet-delivered programs are a valid alternative to face-to-face treatments. Aim of this project to assess the effectivity of two eight-week online-programs consisting of cognitive-behavioral (COPE) and mindfulness-based (MIND) interventions for women with HSDD. Both treatments will be compared to a waitlist-control group. For this project, two well-established group-treatment manuals will be translated into German and adapted to a multimedia online-environment. All participants will be guided through the programs by well-qualified eCoaches.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* female gender
* able to read, write and speak German
* Meet criteria of ICD-10 criteria of Hypoactive Sexual Desire Disorder (established via online-screening and telephone interview)
* Experience significant sexuality-related personal distress (established via online-screening and telephone interview)

Exclusion Criteria:

* currently pregnant
* ongoing medical or psychological treatment for low desire or other sexual dysfunctions or plans to enter such treatment (e.g., in-person sexual therapy, couples therapy) during study participation
* suicide ideation (established via telephone interview)
* currently experiencing significant symptoms of a mental disorder that might interfere with study participation (e.g., Eating Disorders, Obsessive-Compulsive Disorder, Posttraumatic Stress Disorder, Major Depression, Bipolar Disorder) as established via telephone interview
* currently experiencing significant symptoms of a physical condition that might interfere with study participation (e.g., cancer, multiple sclerosis) as established via telephone interview
* current Substance-Abuse Disorder
* current or lifetime Psychotic Disorder
* significant relationship discord or violence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Sexual Interest and Desire Inventory Female (SIDI-F) | at baseline, 5 weeks after baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  The SIDI-F is a clinician-rated instrument consisting of 13 items designed to assess HSDD severity in women. A self-report version, modified for the use in partnered and unpartnered women will be applied.

SECONDARY OUTCOMES:
Female Sexual Distress Scale Revised (FSDS-R) | at baseline, 5 weeks after baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  The Female Sexual Distress Scale (FSDS) is a 13-item self- assessment questionnaire for the evaluation of sexually related personal distress.

OTHER OUTCOMES:
Desire subscale of the Female Sexual Function Index | at baseline, 5 weeks after baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  The Female Sexual Function Index measures women's sexual function with 19-items. Here, the two items assessing sexual desire will be used.
Patient Health Questionnaire 9 (PHQ-9) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 9-item self-report measure used to assess symptoms of depression.
Generalized Anxiety Disorder 7 (GAD-7) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 7-item self-report measure used to assess symptoms of anxiety.
Scale of Body Connection (SBC) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 20-item self-report measure used to assess body awareness
Mindful Attention and Awareness Scale (MAAS) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 15-item self-report measure used to assess mindfulness
Body Image Self-Consciousness Scale | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 15-item self-report measure used to assess body-related self-consciousness
Self-Compassion Scale (SCS) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 12-item self-report scale used to assess self-compassion.
Rumination-Reflection Questionnaire - Adapted Rumination Subscale (RRQ) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  A 12-item scale that assess rumination about sexual issues
Health Action Process Approach (HAPA) | at baseline, 3 months after baseline, 6 months after baseline, 12 months after baseline
  Treatment adherence as measured with the HAPA scales
Working alliance inventory (WAI) adapted for online treatments | 3 months after baseline, 6 months after baseline
  Measures working alliance with eCoaches and online-program
Inventory for the Assessment of Negative Effects of Psychotherapy (INEP) | 3 months after baseline, 6 months after baseline
  15-item self-report measure that assesses side-effects of psychological treatments
Client Satisfaction Questionnaire (CSQ-8) | 3 months after baseline, 6 months after baseline, 12 months after baseline
  8-item self-report measure that assesses women's satisfaction with the online treatment they received
Single target implicit association task (ST-IAT) | at baseline, 3 months after baseline
  An experimental paradigm used to assess implicit cognitive biases towards sexual stimuli
Scrambled-sentences task | at baseline, 3 months after baseline
  An experimental paradigm used to assess implicit cognitive biases towards sexual stimuli
Qualitative evaluation of COPE and MIND | 12 weeks after baseline
  Qualitative telephone interviews with approx. 50 participants to assess perceived mechanisms of change as well as strengths and weaknesses of the programs

CONTACTS AND LOCATIONS:
Overall Officials: Julia Velten, PhD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD data of accepted publications will be published open access on the respective Journal's website or on the Open Science Framework.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Velten J, Hirschfeld G, Meyers M, Margraf J. Results of a randomized waitlist-controlled trial of online cognitive behavioral sex therapy and online mindfulness-based sex therapy for hypoactive sexual desire dysfunction in women. J Consult Clin Psychol. 2024 Nov;92(11):742-755. doi: 10.1037/ccp0000922. Epub 2024 Oct 24. PMID 39446648
- [Derived] Meyers M, Margraf J, Velten J. Psychological Treatment of Low Sexual Desire in Women: Protocol for a Randomized, Waitlist-Controlled Trial of Internet-Based Cognitive Behavioral and Mindfulness-Based Treatments. JMIR Res Protoc. 2020 Sep 29;9(9):e20326. doi: 10.2196/20326. PMID 32990248